CLINICAL TRIAL: NCT04297540
Title: Neuromodulation Technique for the Rehabilitation of Social Skills in Childhood Ataxia
Brief Title: Neuromodulation of Social Skills in Childhood Ataxia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 742
Record Dates: First submitted 2020-02-24; First posted 2020-03-05 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Ataxia, Cerebellar
Keywords: transcranial direct current stimulation; Childhood ataxia; cerebellum; social skills; virtual reality
MeSH Terms: conditions — Cerebellar Ataxia; Social Skills

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active-tDCS group (Experimental): 8 sessions (in two weeks) of active tDCS combined with a virtual reality training
  Interventions: Device: Active-tDCS group
- Sham-tDCS group (Sham Comparator): 8 sessions (in two weeks) of sham tDCS combined with a virtual reality training
  Interventions: Device: Sham-tDCS group

INTERVENTIONS:
Device: Active-tDCS group — Active anodal-tDCS will be delivered over the cerebellum for 8 sessions in two weeks. tDCS will be delivered via a battery driven direct current stimulator. Saline-soaked sponges electrodes will be placed on the cerebellar vermis (anodal electrode) and over the right buccinator muscle (reference electrode). Stimulation intensity will be set at 1.5 mA. The intensity of the stimulation will be gradually increase in order to reach the 1.5 mA with a ramping-up phase of 15 sec. Similarly, a ramping-down phase of 15 sec will gradually decrease the intensity before the end of the stimulation. The duration of the 1.5mA stimulation will be 20 minutes. Soon after the end of the stimulation, the virtual reality training will be performed. The virtual reality training will took place in a child-friendly scenario. It will comprise a total of 80 trials, during which participants will be asked to compete with some avatars in order to activate and to win some objects.
  Arms: Active-tDCS group
Device: Sham-tDCS group — Sham -tDCS will be delivered over the cerebellum for 8 sessions in two weeks. tDCS will be delivered via a battery driven direct current stimulator. Saline-soaked sponges electrodes will be placed on the cerebellar vermis (anodal electrode) and over the right buccinator muscle (reference electrode). Stimulation intensity will be set at 1.5 mA but the current will be applied for 30 sec. The intensity of the stimulation will be gradually increase in order to reach the 1.5 mA with a ramping-up phase of 15 sec. Similarly, a ramping-down phase of 15 sec will gradually decrease the intensity before the end of the stimulation. The duration of the 0mA stimulation will be 20 minutes. Soon after the end of the stimulation, the virtual reality training will be performed. The virtual reality training will took place in a child-friendly scenario. It will comprise a total of 80 trials, during which participants will be asked to compete with some avatars in order to activate and to win some objects.
  Arms: Sham-tDCS group

SUMMARY:
The present study aims to define a protocol of electrical stimulation of the cerebellum via transcranial direct current stimulation (tDCS) combined with a virtual reality protocol to assist the rehabilitation of social skills in adolescents and young adults with childhood ataxia.

Taking into account the high neuronal density of the cerebellum, its strong connection with the cerebral cortex, and its involvement in motor, cognitive and affective processes, as well its involvement in social prediction abilities, the investigators hypothesized that excitatory stimulation of the cerebellum might improve social prediction abilities in adolescents and young adults with childhood ataxia. Moreover, as suggested by previous studies investigating the effect of tDCS in paediatric population, the investigators expected that tDCS will be safe and well tolerated. Such a result would encourage the use of non-invasive brain stimulation in the rehabilitation of social skills in childhood ataxia.

DETAILED DESCRIPTION:
The investigators planned a single centre, randomized stratified, double-blind, sham- controlled design.

Adolescents and young adults with childhood ataxia will be recruited and randomly assigned to two different groups: the active-tDCS group and the sham-tDCS group. Each group will undergo a multi-sessions (8 sessions) intervention during which tDCS will be delivered over the cerebellum. The stimulation will be paired with a virtual reality VR training. The Virtual Reality (VR) training will exploit a design based on probabilistic learning of social events in child-friendly environments. During the training, participants will be asked to conquer some goal/objects by predicting the behaviour of some competing virtual avatars whose actions should be probabilistically learned. Based on the same structures, two different child-friendly scenarios will be created and they will be respectively used in the pre- and in the post-training evaluation sessions (scenario A) or in association with the tDCS protocol throughout the 8 sessions of intervention (scenario B).

Participants' abilities of social prediction (primary outcome) will be tested through a validated computer based Action prediction task assessing participants' abilities in predicting others' actions based on previous experience. This experimental paradigm comprises a probabilistic learning (familiarization) phase and a testing phase. In the familiarization phase participants are asked to observe an actor performing two different types of grasping actions (such as grasping movement of an apple for eating the apple or for offering the apple to another partner) in different colour-cued contexts. They are asked to recognise actor's intention.

Crucially, the probability of co-occurrence between one action and the colour-cued context is implicitly biased with pre-established probability of association. In the testing phase, the same videos are presented but their length is dramatically shortened via temporal occlusion before the action is completed. In this way, since the movement kinematics is ambiguous, an observer would use the previously learned association with context to predict the fate of the action, and responses should be biased toward the contextual priors. A control non-social prediction task with a similar structure will be also used. A standard neuropsychological assessment (NEPSY-II) before and after the training will allow assessing the generalizability of the effects to general social perception abilities, in particular Theory of Mind and affect recognition (Secondary Outcomes). In the post-training and in the follow-up evaluation session (one month after the end of the intervention) the training acceptability and the quality of life assessments will be performed.

The protocol will allow testing the efficiency of the combined tDCS+ VR training in:

* enhancing social prediction abilities in childhood ataxia;
* enhancing implicit learning abilities, even in non social contexts;
* improving theory of mind abilities;
* improving patients' quality of life;
* further investigating the safety and tolerability of tDCS.

ELIGIBILITY:
Inclusion criteria:

* Adolescents and young adults who aged 11-25 years
* Childhood ataxia
* Intelligence Quotient > 80

Exclusion Criteria:

* Presence of contraindication to tDCS (history of epilepsy, migraine, severe brain trauma; presence of metal in the brain/skull or implanted neurostimulator, cardiac pacemaker; state of pregnancy)
* Intake of or withdrawal from some drugs potentially changing the seizure threshold
* Presence of comorbidity with an important medical conditions
* Severe sensorial, motor and/or behavioural problems that could interfere with the use of GRAIL/VR technology

Ages: 11 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
Change in Social Prediction abilities in the Action Prediction task | Time 1- at the end the last training session vs Time 0- before starting the first training session
  -Performance in the testing phase of the action prediction task, consisting in the accuracy in discriminating between two alternatives in order to predict the unfolding of an individual or interpersonal action as a function of different probability of co-occurence between the same action and a contextual cues, as previously learned during a familiarization phase.
Change in Social Prediction abilities in the Virtual Reality scenario | Time 1- at the end the last training session vs Time 0- before starting the first training session
  -Performance in the evaluation session in the Virtual Reality scenario, consisting in the percentage difference in the objects activated by the participants with respect to the objects activated by the avatars.

SECONDARY OUTCOMES:
Change in Non-social Prediction task abilities | Time 1- at the end the last training session vs Time 0- before starting the first training session
  Performance in the testing phase of the shape prediction task, consisting in the accuracy in discriminating between two alternatives in order to predict the shape of a moving object as a function of different probability of co-occurence between the same shape and a contextual cues, as previously learned during a familiarization phase.
Change in Social Cognition | Time 2- up to one month after the end of the intervention vs Time 0- before starting the first training session
  Theory of Mind Parts A and B and Emotion Recognition of the NEPSY-II testing battery (Scaled scores ranging 1 to 19, mean=10, standard deviation=3, with higher scores meaning better performance).
Change in Quality of life assessment: TNO-AZL Questionnaires for Children's Health-Related Quality of Life (TACQOL) questionnaire | Time 2- up to one month after the end of the intervention vs Time 0- before starting the first training session
  Overall functioning and quality of life assessed using the TNO-AZL Questionnaires for Children's Health-Related Quality of Life (TACQOL), presented in two forms: the self-compiled one and the parent compiled one. The questionnaire comprises 8 different subscales referring to problems/limitations in general physical functioning (Body subscale);.in motor functioning (Motor subscales); in independent daily functioning (Auto subscale); in cognitive functioning and school performance (cognit subscale); in social contacts with parents and peers (Social scale); to the occurrence of positive moods (Empos subscale) or negative moods (Emoneg scale). The sum scores may range from 0 to 32 for Body, Motor, Cognit, Auto and Social scales. For Empos and Emoneg the scores vary between 0 and 16.
  The calculated scale scores are all in the same direction: a low score indicates a lower Health-Related Quality of Life (HRQoL); a high score indicates a higher HRQoL.
training feasibility assessment: Evaluation of the number of dropouts | Time 1- at the end the last training session
  Evaluation of the number of dropouts: number of patient who renounce to complete the whole training Evaluation of the number of sessions completed per patient: total number of sessions performed in front of the total number proposed of eight sessions
training acceptability assessment: Ad-hoc questionnaire | Time 1- at the end the last training session
  Ad-hoc questionnaire completed by participants and by their parents to assess subjective evaluation of training accessibility and efficacy (10 cm Visual Analogue scales with higher values corresponding to greater agreement).